CLINICAL TRIAL: NCT01722422
Title: Hyperoxia and Hypertonic Saline in Septic Shock
Acronym: Hyper2S
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PHRC 11-05
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Septic Shock; Adult Respiratory Distress Syndrome
Keywords: sepsis; shock; hyperoxia; hypertonic saline
MeSH Terms: conditions — Shock, Septic; Respiratory Distress Syndrome; Sepsis; Shock; Hyperoxia | interventions — Oxygen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- normoxia and isotonic saline (Placebo Comparator): Administration of oxygen in order to maintain SaO2 between 88% and 95%. Fluid resuscitation if needed with isotonic saline during 3 days.
  Interventions: Drug: oxygen and saline
- normoxia and 3% hypertonic saline (Active Comparator): Administration of oxygen in order to maintain SaO2 between 88% and 95%. Fluid resuscitation if needed with 3% hypertonic saline during 3 days.
  Interventions: Drug: oxygen and saline
- hyperoxia and isotonic saline (Active Comparator): Administration of oxygen with FiO2 = 100% during the first 24 hours and after switch oxygen administration to usual care.
  Fluid resuscitation if needed with isotonic saline during 3 days.
  Interventions: Drug: oxygen and saline
- hyperoxia and 3% hypertonic saline (Active Comparator): Administration of oxygen with FiO2 = 100% during the first 24 hours and after switch oxygen administration to usual care.
  Fluid resuscitation if needed with 3% hypertonic saline during 3 days.
  Interventions: Drug: oxygen and saline

INTERVENTIONS:
Drug: oxygen and saline

SUMMARY:
Assessment of the effect of hyperoxia and hypertonic saline on survival in patients with septic shock Hyperoxia and hypertonic saline may have beneficial effects on organ perfusion and oxygenation and may reduce the organ failure occurences. To date, only scarce data are available. Side effects are not well described. Therefore we designed a randomized clinical trial in order to assess the early administration of hypertonic saline and oxygen in the very early beginning of septic shock.

DETAILED DESCRIPTION:
The study is designed as factorial 2x2. Patients will be stratified at the randomisation according the presence or absence of Acute Respiratory Distress Syndrome in order to perform a sub group analysis for all outcome criteria.

ELIGIBILITY:
Inclusion Criteria:

* patients with less than 6 hours septic shock according criteria of Bone
* minimal dose of catecholamines at least 0.1 µg/Kg/min
* patient with mechanical ventilation
* written informed consent

Exclusion Criteria:

* age < 18 years
* pregnancy
* participation in other trial with the same endpoint
* moribund
* absence of registration in french health care system
* patient protected by law
* hypernatremia < 130 mmol/l ou > 145 mmol/l
* patient with P/F < 100 mm Hg with PEEP > 5 cms of water
* intracranial hypertension
* patient admitted for cardiac arrest
* overt cardiac failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | day 28

SECONDARY OUTCOMES:
all-cause mortality | day 90
evolution of organ failures | day 1 to day 28
catecholamines free days | day 1 to day 28
mechanical ventilation free days | day 1 to day 28
safety data | day 1 to day 90

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Angers, Angers, France

REFERENCES:
- [Background] Calzia E, Asfar P, Hauser B, Matejovic M, Ballestra C, Radermacher P, Georgieff M. Hyperoxia may be beneficial. Crit Care Med. 2010 Oct;38(10 Suppl):S559-68. doi: 10.1097/CCM.0b013e3181f1fe70. PMID 21164398
- [Background] Goertz AW, Mehl T, Lindner KH, Rockemann MG, Schirmer U, Schwilk B, Georgieff M. Effect of 7.2% hypertonic saline/6% hetastarch on left ventricular contractility in anesthetized humans. Anesthesiology. 1995 Jun;82(6):1389-95. doi: 10.1097/00000542-199506000-00010. PMID 7540812
- [Background] Oliveira RP, Weingartner R, Ribas EO, Moraes RS, Friedman G. Acute haemodynamic effects of a hypertonic saline/dextran solution in stable patients with severe sepsis. Intensive Care Med. 2002 Nov;28(11):1574-81. doi: 10.1007/s00134-002-1509-x. Epub 2002 Oct 1. PMID 12415443
- [Background] Junger WG, Hoyt DB, Davis RE, Herdon-Remelius C, Namiki S, Junger H, Loomis W, Altman A. Hypertonicity regulates the function of human neutrophils by modulating chemoattractant receptor signaling and activating mitogen-activated protein kinase p38. J Clin Invest. 1998 Jun 15;101(12):2768-79. doi: 10.1172/JCI1354. PMID 9637711
- [Background] Coimbra R, Hoyt DB, Junger WG, Angle N, Wolf P, Loomis W, Evers MF. Hypertonic saline resuscitation decreases susceptibility to sepsis after hemorrhagic shock. J Trauma. 1997 Apr;42(4):602-6; discussion 606-7. doi: 10.1097/00005373-199704000-00004. PMID 9137245
- [Derived] Commereuc M, Nevoret C, Radermacher P, Katsahian S, Asfar P, Schortgen F; HYPER2S investigators. Hyperchloremia is not associated with AKI or death in septic shock patients: results of a post hoc analysis of the "HYPER2S" trial. Ann Intensive Care. 2019 Aug 22;9(1):95. doi: 10.1186/s13613-019-0570-3. PMID 31440853
- [Derived] Asfar P, Schortgen F, Boisrame-Helms J, Charpentier J, Guerot E, Megarbane B, Grimaldi D, Grelon F, Anguel N, Lasocki S, Henry-Lagarrigue M, Gonzalez F, Legay F, Guitton C, Schenck M, Doise JM, Devaquet J, Van Der Linden T, Chatellier D, Rigaud JP, Dellamonica J, Tamion F, Meziani F, Mercat A, Dreyfuss D, Seegers V, Radermacher P; HYPER2S Investigators; REVA research network. Hyperoxia and hypertonic saline in patients with septic shock (HYPERS2S): a two-by-two factorial, multicentre, randomised, clinical trial. Lancet Respir Med. 2017 Mar;5(3):180-190. doi: 10.1016/S2213-2600(17)30046-2. Epub 2017 Feb 15. PMID 28219612